CLINICAL TRIAL: NCT00556673
Title: An Exploratory, Multi-centre, Double-blind, Placebocontrolled Crossover Study, to Investigate the Bronchodilatory Efficacy of a Single Dose of Indacaterol in Fixed Combination With Mometasone Furoate Delivered Via a MDDPI (Twisthaler®) in Adult Patients With Persistent Asthma Using Open Label Seretide® Accuhaler® (50/250 Mcg b.i.d.) as an Active Control
Brief Title: Bronchodilatory Efficacy of a Single Dose QMF149 (Indacaterol Maleate/Mometasone Furoate) Via the Twisthaler® Device in Adult Patients With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQMF149A2204; 2007-002360-10 (EudraCT Number)
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-03

CONDITIONS: Asthma
Keywords: Asthma, QMF149, fixed combination of indacaterol and mometasone furoate
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; QMF149; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indacaterol/mometasone - Placebo (Experimental): In Treatment Period 1 (Day 1) participants received 2 inhalations of indacaterol maleate 250 μg / mometasone furoate 200 μg once a day in the morning via the Twisthaler device. In Treatment Period 2 (Day 8) participants received 2 inhalations of placebo via the Twisthaler device once a day in the morning. In Treatment Period 3 (Day 15) participants received fluticasone proprionate 250 μg / salmeterol xinafoate 50 μg twice a day delivered via dry-powder inhaler. Each treatment period was separated by a minimum washout period of 7 days.
  Interventions: Drug: indacaterol maleate/mometasone furoate; Drug: placebo to indacaterol maleate/mometasone furoate; Drug: fluticasone proprionate / salmeterol xinafoate
- Placebo - indacaterol/mometasone (Experimental): In Treatment Period 1 (Day 1) participants received 2 inhalations of placebo in the morning via the Twistheler device. In Treatment Period 2 (Day 8) participants received 2 inhalations of indacaterol maleate 250 μg / mometasone furoate 200 μg via the Twisthaler device in the morning. In Treatment Period 3 (Day 15) participants received fluticasone proprionate 250 μg / salmeterol xinafoate 50 μg twice a day delivered via dry-powder inhaler. Each treatment period was separated by a minimum washout period of 7 days.
  Interventions: Drug: indacaterol maleate/mometasone furoate; Drug: placebo to indacaterol maleate/mometasone furoate; Drug: fluticasone proprionate / salmeterol xinafoate

INTERVENTIONS:
Drug: indacaterol maleate/mometasone furoate — Indacaterol maleate 250 μg / mometasone furoate 200 μg delivered via the Twisthaler device.
  Other Names: QMF149
Drug: placebo to indacaterol maleate/mometasone furoate — Placebo to indacaterol maleate/mometasone furoate delivered via the Twisthaler device.
Drug: fluticasone proprionate / salmeterol xinafoate — Fluticasone proprionate 250 μg / salmeterol xinafoate 50 μg delivered via the Accuhaler® device.
  Other Names: Seretide® Accuhaler®

SUMMARY:
This study is designed to evaluate the bronchodilatory efficacy of indacaterol maleate 500 μg/mometasone furoate 400 μg via the Twisthaler® device in adult patients with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients aged 18-75 years with persistent asthma
* Patients with persistent asthma, diagnosed according to the Global Initiative for Asthma guidelines (GINA) and who additionally met the following criteria:

  1. Patients receiving daily treatment with inhaled corticosteroid up to the maximum dose per day indicated in the package leaflet, in a stable regimen for the month prior to Visit 1.
  2. Patients with a forced expiratory volume in 1 second (FEV1) at Visit 1 of ≥ 50% of the predicted normal value. This criterion for FEV1 had to be demonstrated after a washout period of at least 6 hours during which no short acting β2-agonist had been inhaled, and a minimum of 48 hours for a long acting β2-agonist.
  3. Patients who demonstrated an increase of ≥12% and ≥200 mL in FEV1 over their pre-bronchodilator value 30 minutes after inhaling a total of 200 μg of salbutamol (or albuterol) via metered dose inhaler (MDI) (the reversibility test). Reversibility had to be demonstrated after an appropriate washout period of at least 6 hrs prior to the evaluation for a shortacting β2-agonist. The administration of salbutamol (or albuterol) for the reversibility test was to be within 30 minutes after pre-bronchodilator spirometry. Reversibility had to be demonstrated at Visit 1 or between Visits 1 and 2, in order for patients to be included in the trial.
  4. For each patient, the smaller value of the Visit 1 FEV1 or the Visit 2 FEV1 pre-dose value had to be at least 85% of the larger value.
* Body mass index (BMI) between 18 and 32 kg/m^2 and weight >50 kg.
* patients using local contraception

Exclusion Criteria:

* Pregnant or nursing women
* Recent use of tobacco or history of smoking > 10 pack years
* Patients diagnosed with chronic obstructive pulmonary disease (COPD)
* Patients with recent experience of severe asthma attack/exacerbation within 6-months of study start
* Patients with frequent rescue medication (>8 puffs/day for two consecutive days)
* Clinically relevant laboratory abnormality or a clinically significant condition
* Active cancer or a history of cancer with less than 5 years disease free survival time
* History of long QT syndrome or with long QTc interval prior to dosing
* History of hypersensitivity to the study drugs or to drugs with similar chemical structures
* Use of certain medications
* Use of other investigational drugs
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result
* History of immunodeficiency diseases, including a positive human immumodeficiency virus (HIV) test result.
* History of drug or alcohol abuse or evidence of such abuse

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (2):
- Novartis Investigator Site, Poitiers, France
- Novartis Investigator Site, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Indacaterol/Mometasone - Placebo: In Treatment Period 1 (Day 1) participants received 2 inhalations of indacaterol maleate 250 μg/mometasone furoate 200 μg once a day in the morning via the Twisthaler device. In Treatment Period 2 (Day 8) participants received 2 inhalations of placebo via the Twisthaler device once a day in the morning. In Treatment Period 3 (Day 15) participants received fluticasone proprionate 250 μg/salmeterol xinafoate 50 μg twice a day delivered via dry-powder inhaler. Each treatment period was separated by a minimum washout period of 7 days.
- Placebo - Indacaterol/Mometasone: In Treatment Period 1 (Day 1) participants received 2 inhalations of placebo in the morning via the Twisthaler device. In Treatment Period 2 (Day 8) participants received 2 inhalations of indacaterol maleate 250 μg/mometasone furoate 200 μg via the Twisthaler device in the morning. In Treatment Period 3 (Day 15) participants received fluticasone proprionate 250 μg/salmeterol xinafoate 50 μg twice a day delivered via dry-powder inhaler. Each treatment period was separated by a minimum washout period of 7 days.
Period: Overall Study
Arm/Group | Indacaterol/Mometasone - Placebo | Placebo - Indacaterol/Mometasone
Started | 16 | 15
Pharmacodynamic (PD) Population | 12 (4 patients inadvertently unblinded were not included in PD analysis population.) | 12 (3 patients inadvertently unblinded were not included in PD analysis population.)
Completed | 13 | 13
Not Completed | 3 | 2
Not completed — Protocol deviation | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol/Mometasone - Placebo | Placebo - Indacaterol/Mometasone | Total
Number analyzed (Participants) | 16 | 15 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 39.1 (11.93) | 41.5 (7.23) | 40.3 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Period Baseline to 24 Hour Post-dose (Trough) Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Change from the period baseline to 24 hour post dose trough FEV1 after 1 day of treatment was modeled using a linear mixed effect model fitting treatment, sequence and period as fixed factors, patient within sequence as a random factor and pre-dose FEV1 as covariate.
Time Frame: Pre-dose for each Treatment Period (Days 1, 8 and 15) and 24-hours post-dose for each Treatment Period (Days 2, 9 and 16).
Population: Pharmacodynamic population included all patients randomized that received at least one dose of study drug and completed the first two treatment periods with evaluable data for the primary efficacy variable, and with no major protocol deviations. 7 patients who were inadvertently unblinded by the investigator were excluded from the PD analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: liters
Groups:
- Indacaterol/Mometasone: Participants received a single dose of indacaterol/mometasone 500/400 μg delivered via the TWISTHALER device (2 inhalations of 250/200 μg) in the morning.
- Placebo: Participants received 2 inhalations of placebo to indacaterol/mometasone via the TWISTHALER device in the morning.
- Fluticasone/Salmeterol: Participants received fluticasone/salmeterol 250/50 μg via dry powder inhaler (DPI), one inhalation in the morning and one inhalation the following evening.
Arm/Group | Indacaterol/Mometasone | Placebo | Fluticasone/Salmeterol
Number analyzed (Participants) | 24 | 24 | 24
liters | 0.27 [0.19 to 0.36] | -0.12 [-0.21 to -0.04] | 0.37 [0.28 to 0.47]
Statistical Analysis 1: Comparison: Indacaterol/Mometasone vs Placebo; The primary hypothesis tested was that the change from period baseline of trough FEV1 for placebo and indacaterol/mometasone was equal. The one-sided alternative was that the increase from period baseline of trough FEV1 for indacaterol/mometasone was higher than for placebo; Test type: Superiority or Other; p < 0.0001, 1-sided — Linear mixed effect model fitting treatment, sequence and period as fixed factors, patient within sequence as a random factor and pre-dose FEV1 as covariate. A significance level of 5% was used to determine statistical significance; LS Mean Difference = 0.39, 90% CI 2-sided [0.28 to 0.51]

2. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Peak FEV1 is defined as the peak FEV1 between 0 and 4 hours post-dose. The change from baseline in peak FEV1 was modeled using a linear mixed effect model fitting treatment, sequence and period as fixed factors, patient within sequence as a random factor and pre-dose FEV1 as covariate.
Time Frame: Days 1, 8 and 15, pre-dose (Baseline) and 5, 15, and 30 minutes, 1, 2, 3, and 4 hours post-dose.
Population: Pharmacodynamic population
Measure: Least Squares Mean (90% Confidence Interval); unit: liters
Arm/Group | Indacaterol/Mometasone | Placebo | Fluticasone/Salmeterol
Number analyzed (Participants) | 24 | 24 | 24
liters | 0.64 [0.55 to 0.73] | 0.26 [0.17 to 0.34] | 0.62 [0.54 to 0.71]

3. Secondary Outcome: Change From Period Baseline in Trough Percent Predicted Forced Expiratory Volume in 1 Second (FEV1)
Description: Trough FEV1 was measured 24 hours post-dose. The FEV1 percent predicted expresses FEV1 as a percentage of the "predicted values" for participants of similar characteristics (height, age, sex, and sometimes race and weight). A positive change from baseline in FEV1 % predicted indicates improvement in lung function. Change from baseline in trough FEV1 % predicted was modeled using a linear mixed effect model fitting treatment, sequence and period as fixed factors, patient within sequence as a random factor and pre-dose value as covariate.
Time Frame: as for outcome 1
Population: Pharmacodynamic population
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent of predicted
Arm/Group | Indacaterol/Mometasone | Placebo | Fluticasone/Salmeterol
Number analyzed (Participants) | 24 | 24 | 24
Percent of predicted | 6.95 [4.68 to 9.22] | -2.87 [-5.14 to -0.59] | 9.85 [7.58 to 12.12]

4. Secondary Outcome: Change From Period Baseline in Peak Percent Predicted Forced Expiratory Volume in 1 Second (FEV1)
Description: Peak FEV1 was defined as the peak FEV1 up to 4 hours post-dose. The FEV1 percent predicted expresses FEV1 as a percentage of the "predicted values" for participants of similar characteristics (height, age, sex, and sometimes race and weight). A positive change from baseline in FEV1 % predicted indicates improvement in lung function. Change from baseline in peak FEV1 % predicted was modeled using a linear mixed effect model fitting treatment, sequence and period as fixed factors, patient within sequence as a random factor and pre-dose value as covariate.
Time Frame: Days 1, 8 and 15, pre-dose (Baseline) and 5, 15, and 30 minutes, 1, 2, 3, and 4 hours post-dose.
Population: Pharmacodynamic population
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent of predicted
Arm/Group | Indacaterol/Mometasone | Placebo | Fluticasone/Salmeterol
Number analyzed (Participants) | 24 | 24 | 24
Percent of predicted | 16.27 [14.24 to 18.29] | 6.85 [4.83 to 8.88] | 16.49 [14.47 to 18.51]

5. Secondary Outcome: Change From Period Baseline in Trough Forced Vital Capacity (FVC)
Description: Vital capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Trough FVC was measured 24 hours post-dose. Change form baseline in trough FVC was modeled using a linear mixed effect model fitting treatment, sequence and period as fixed factors, patient within sequence as a random factor and pre-dose value as covariate.
Time Frame: as for outcome 1
Population: Pharmacodynamic population
Measure: Least Squares Mean (90% Confidence Interval); unit: liters
Arm/Group | Indacaterol/Mometasone | Placebo | Fluticasone/Salmeterol
Number analyzed (Participants) | 24 | 24 | 24
liters | 0.22 [0.13 to 0.31] | -0.14 [-0.23 to -0.05] | 0.17 [0.08 to 0.27]

6. Secondary Outcome: Change From Period Baseline in Peak Forced Vital Capacity (FVC)
Description: Vital capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Peak FVC was measured up to 4 hours post-dose. Change from baseline in peak FVC was modeled using a linear mixed effect model fitting treatment, sequence and period as fixed factors, patient within sequence as a random factor and pre-dose value as covariate.
Time Frame: Days 1, 8 and 15, pre-dose (Baseline) and 5, 15, and 30 minutes, 1, 2, 3, and 4 hours post-dose.
Population: Pharmacodynamic population
Measure: Least Squares Mean (90% Confidence Interval); unit: liters
Arm/Group | Indacaterol/Mometasone | Placebo | Fluticasone/Salmeterol
Number analyzed (Participants) | 24 | 24 | 24
liters | 0.47 [0.38 to 0.55] | 0.20 [0.12 to 0.29] | 0.35 [0.27 to 0.44]

7. Secondary Outcome: Change From Period Baseline in Trough FEV1/FVC Ratio
Description: The forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) ratio represents the proportion of a person's vital capacity that they are able to expire in the first second of an expiration. Trough FEV1/FVC was calculated from measurements taken 24 hours post-dose. Change from baseline in trough FEV1/FVC ratio was modeled using a linear mixed effect model fitting treatment, sequence and period as fixed factors, patient within sequence as a random factor and pre-dose value as covariate.
Time Frame: as for outcome 1
Population: Pharmacodynamic population
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Indacaterol/Mometasone | Placebo | Fluticasone/Salmeterol
Number analyzed (Participants) | 24 | 24 | 24
ratio | 2.50 [2.28 to 2.72] | 2.15 [1.93 to 2.37] | 2.65 [2.43 to 2.87]

8. Secondary Outcome: Change From Period Baseline in Peak FEV1/FVC Ratio
Description: The forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) ratio represents the proportion of a person's vital capacity that they are able to expire in the first second of an expiration. Peak FEV1/FVC was calculated from spirometry measurements taken up to 4 hours post-dose. Change from baseline in peak FEV1/FVC ratio was modeled using a linear mixed effect model fitting treatment, sequence and period as fixed factors, patient within sequence as a random factor and pre-dose value as covariate.
Time Frame: Days 1, 8 and 15, pre-dose (Baseline) and 5, 15, and 30 minutes, 1, 2, 3, and 4 hours post-dose.
Population: Pharmacodynamic population
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Indacaterol/Mometasone | Placebo | Fluticasone/Salmeterol
Number analyzed (Participants) | 24 | 24 | 24
ratio | 2.86 [2.63 to 3.10] | 2.53 [2.30 to 2.76] | 2.90 [2.67 to 3.14]

9. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 12 Hours Post-dose for Mometasone Furoate
Time Frame: Samples were taken pre-dose and at 15 and 30 minutes and 1, 2, 4, and 12 hours post-dose.
Population: All participants with evaluable pharmacokinetic (PK) parameter data were included in the PK data analysis.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Indacaterol/Mometasone
Number analyzed (Participants) | 29
pg*h/mL | 287 (140)

10. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 Hours Post-dose for Mometasone Furoate
Time Frame: Samples were taken pre-dose and at 15 and 30 minutes and 1, 2, 4, 12 and 24 hours post-dose.
Population: All participants with evaluable pharmacokinetic (PK) parameter data were included in the PK data analysis.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Indacaterol/Mometasone
Number analyzed (Participants) | 29
pg*h/mL | 389 (191)

11. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 Hours Post-dose for Indacaterol
Time Frame: Samples were taken pre-dose and at 15 and 30 minutes and 1, 2, 4, 12 and 24 hours post-dose.
Population: All participants with evaluable pharmacokinetic (PK) parameter data were included in the PK data analysis.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Indacaterol/Mometasone
Number analyzed (Participants) | 28
pg*h/mL | 1331 (712)

12. Secondary Outcome: Maximum (Peak) Plasma Concentration (Cmax) of Mometasone Furoate
Time Frame: Samples were taken pre-dose and at 15 and 30 minutes and 1, 2, 4, 12 and 24 hours post-dose.
Population: All participants with evaluable pharmacokinetic (PK) parameter data were included in the PK data analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Indacaterol/Mometasone
Number analyzed (Participants) | 29
pg/mL | 47.3 (20.9)

13. Secondary Outcome: Maximum (Peak) Plasma Concentration (Cmax) of Indacaterol
Time Frame: Samples were taken pre-dose and at 15 and 30 minutes and 1, 2, 4, 12 and 24 hours post-dose.
Population: All participants with evaluable pharmacokinetic (PK) parameter data were included in the PK data analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Indacaterol/Mometasone
Number analyzed (Participants) | 28
pg/mL | 289 (133)

14. Secondary Outcome: Time to Reach Peak or Maximum Concentration Following Drug Administration for Mometasone Furoate
Time Frame: Samples were taken pre-dose and at 15 and 30 minutes and 1, 2, 4, 12 and 24 hours post-dose.
Population: All participants with evaluable pharmacokinetic (PK) parameter data were included in the PK data analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Indacaterol/Mometasone
Number analyzed (Participants) | 29
hours | 1.05 [0.250 to 2.08]

15. Secondary Outcome: Time to Reach Peak or Maximum Concentration Following Drug Administration for Indacaterol
Time Frame: Samples were taken pre-dose and at 15 and 30 minutes and 1, 2, 4, 12 and 24 hours post-dose.
Population: All participants with evaluable pharmacokinetic (PK) parameter data were included in the PK data analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Indacaterol/Mometasone
Number analyzed (Participants) | 28
hours | 0.325 [0.267 to 0.617]

ADVERSE EVENTS:
Arm/Group | Indacaterol/Mometasone | Placebo | Fluticasone/Salmeterol
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 10/29 | 6/28 | 2/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol/Mometasone (N=29) | Placebo (N=28) | Fluticasone/Salmeterol (N=26)
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 1 | 1 | 0
Catheter site haematoma (General disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 3 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Premenstrual syndrome (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.